CLINICAL TRIAL: NCT00153179
Title: The Impact of Free Fatty Acid Reduction on Vascular Function and Skeletal Muscle Glucose Utilization in Type 2 Diabetes Mellitus
Brief Title: Free Fatty Acids and Vascular Function in Subjects With Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005P-000088
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance; insulin signaling; endothelium-dependent vasodilation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Acipimox treatment for 7 days
  Interventions: Drug: acipimox
- 2 (Placebo Comparator): placebo treatment for 7 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acipimox — subjects will receive acipimox 250 mg orally every 6 hours (or matching placebo) for 7 days, including a dose at 6am on the morning of the study testing visit
  Other Names: Olbetam
  Arms: 1
Drug: placebo — matching placebo
  Arms: 2

SUMMARY:
This study will test the hypothesis that reduction in release of free fatty acids from adipocytes will restore insulin-mediated endothelium-dependent vasodilation and skeletal muscle glucose metabolism in subject with type 2 diabetes.

DETAILED DESCRIPTION:
During the past two decades, there has been a steady increase in the incidence of diabetes mellitus, such that nearly 17 million people are now afflicted. The vast majority of these have type 2 diabetes. Over the next 40 years, the type 2 diabetic population in the United States is expected to increase to nearly 30 million.

Diabetes substantially increases the risk of atherosclerosis, and thereby, cardiovascular morbidity and mortality. Indeed, cardiovascular disease causes more than 50% of the mortality in patients with diabetes. People with type 2 diabetes manifest two cardinal signs of dysmetabolism: hyperglycemia and insulin resistance. Insulin resistance is a progressive phenomenon that occurs well before the onset of frank diabetes, and results in alterations in insulin signaling. Experimental studies suggest that insulin signaling is required for vascular homeostasis, and its impairment is associated with endothelial dysfunction. In the clinical setting, insulin resistance is associated with atherosclerosis and predicts cardiovascular events independent of hyperglycemia. Therefore, we will study the importance of insulin signaling in endothelial biology in humans and the effects of free fatty acids on endothelial function in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus (as defined by the National Diabetes Data Group)
* normal cardiovascular exam
* non smoker (for 1 year prior to entry)
* Healthy volunteers
* no known medical problems
* normal cardiovascular exam
* fasting glucose < 110 mg/dL
* non-smoker (for 1 year prior to entry)

Exclusion Criteria:

Type 2 Diabetics

* untreated hypertension (>140/90 mmHg)
* untreated hypercholesterolemia (LDL > 75th percentile for age)
* cigarette smoking within 1 year
* neuropathy requiring medication
* nephropathy (> 300mg/24 hour urinary albumin, or serum creatinine > 1.4 mg/dL
* abnormal cardiovascular exam
* treatment with thiazolidinedione within 1 year
* post-menopausal women taking hormone replacement therapy

(Note: subjects taking angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) must stop these medications for 2 weeks prior to taking study drug. If blood pressure rises to >140/90, subjects will be prescribed an alternative medication or be withdrawn from the study.

Healthy Volunteers

* abnormal cardiovascular exam
* use of prescription medications
* fasting glucose > 110mg/dL
* cigarette smoking within 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Creager, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls, Placebo First, Then Acipimox; Healthy Controls, Acipimox First, Then Placebo; Metabolic Syndrome, Placebo First, Then Acipimox; Metabolic Syndrome, Acipimox First, Then Placebo: The study is a randomized, placebo-controlled, double-blind, cross-over trial in subjects with the metabolic syndrome and healthy subjects with interventions assessed over one day of treatment and a washout period of 4 weeks. Acipimox (Pharmacia and Upjohn (Pfizer), Kalamazoo, MI), 250 mg, or matching placebo will be given at 7 PM, 1 AM, and 7 AM, and 11 AM prior to and on the day of study.
Period: Study Visit Day 1
Arm/Group | Healthy Controls, Placebo First, Then Acipimox | Healthy Controls, Acipimox First, Then Placebo | Metabolic Syndrome, Placebo First, Then Acipimox | Metabolic Syndrome, Acipimox First, Then Placebo
Started | 10 | 8 | 13 | 9
Completed | 10 | 8 | 13 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Study Visit Day 2
Arm/Group | Healthy Controls, Placebo First, Then Acipimox | Healthy Controls, Acipimox First, Then Placebo | Metabolic Syndrome, Placebo First, Then Acipimox | Metabolic Syndrome, Acipimox First, Then Placebo
Started | 10 | 8 | 13 | 9
Completed | 9 | 8 | 11 | 7
Not Completed | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Metabolic Syndrome | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 22 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (5.6) | 58.6 (8.1) | 55.6 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation After Placebo or Acipimox Treatment Between Healthy Controls and Those With Metabolic Syndrome
Description: Flow mediated dilation is calculated as follows: A resting arterial diameter measurement is obtained using the average of 10 EKG-gated ultrasound images. Next, an occlusive pressure is applied (using a blood pressure cuff inflated to a suprasystolic pressure)for a period of 5 minutes. After 5 minutes, the cuff is rapidly deflated. This produces a reactive hyperemic response which is captured via ultrasound at 1 minute post cuff deflation (also 10 EKG-gated images averaged). The diameter of the artery following reactive hyperemia is calculated and compared to the resting diameter to obtain a percent dilation. This is flow-mediated dilation.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Flow mediated dilation
Arm/Group | Healthy Controls, Placebo Treatment | Healthy Controls, Acipimox Treatment | Metabolic Syndrome, Placebo Treatment | Metabolic Syndrome, Acipimox Treatment
Number analyzed (Participants) | 17 | 17 | 18 | 18
Flow mediated dilation | 10.65 (4.73) | 11.57 (5.72) | 8.79 (6.90) | 9.52 (6.38)

2. Primary Outcome: Difference in Insulin-mediated Skeletal Muscle Glucose Utilization Between Test Agent and Placebo
Description: Insulin sensitivity (M) is measured by using a hyperinsulinaemic-euglycaemic clamp. Insulin sensitivity (M) was calculated as the average glucose infusion rate (mg/kg of body weight per min) over the last 30 min of the clamp. Higher values indicate better outcomes (more insulin sensitive), while lower values indicate more insulin resistance.
Time Frame: baseline, 7 days
Population: The data for this outcome measure was lost when the investigator left the institution, so the measure was not analyzed.
Arm/Group | Healthy Controls, Placebo Treatment | Healthy Controls, Acipimox Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Healthy Controls: Healthy subjects will be ≥18 years of age and have no known medical problems, have a normal cardiovascular exam and a fasting glucose <110 mg/dL determined during a screening visit.
- Metabolic Syndrome: The patient population for this specific aim will include non-diabetic subjects with the metabolic syndrome who are ≥18 years of age. The metabolic syndrome will be defined as the presence of 4 or 5 components of the syndrome as defined by the National Cholesterol Education Program including abdominal obesity, elevated fasting blood sugar (110 mg/dL< glucose < 126 mg/dL) (54), low HDL, elevated fasting blood triglycerides (Trigs > 150 mg/dL), and hypertension (BP > 140/90 mm HG) (55). Patients will be excluded from this protocol if they have any of the following: diabetes mellitus, untreated hypercholesterolemia (LDL > 75th percentile for age), cigarette smoking within 1 year, renal insufficiency (creatinine > 1.4 mg/dl), blood dyscrasia, or hepatic dysfunction (ALT > 2x normal). Potential subjects will also be excluded if they are infected with the human immunodeficiency virus or have psychiatric illness requiring more than one medication for depression or anxiety.
Arm/Group | Healthy Controls | Metabolic Syndrome
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No